CLINICAL TRIAL: NCT00642785
Title: A Research Study Examining the Effectiveness of Distant Activation of ACE Pigments Associated With Recurrent Human Herpes Simplex Virus-Induced Skin Lesions.
Brief Title: Activation of Alternative Cellular Energy (ACE) Pathway in the Therapy of Herpes Virus Infections
Status: Completed | Type: Observational
Sponsor: Institute of Progressive Medicine (Other)
Responsible Party: W. John Martin, Medical Director, Institute of Progressive Medicine
Other Study IDs: 071/081
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Herpes Simplex; Herpes Zoster
Keywords: herpes; HSV; zoster; HZV; shingles
MeSH Terms: conditions — Herpes Simplex; Herpes Zoster

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Patients with active oral or genital HSV skin lesions
- 2: Patients with a history of recurrent oral or genital HSV but without an active lesion at the time of treatment
- 3: Patients with active shingles/zoster
- 4: Patients with post herpetic neuralgia

SUMMARY:
The research question to be addressed is whether indirect phototherapy based activation of the body's alternative cellular energy (ACE) pathway will lead to expedited healing of active herpes simplex virus (HSV) and herpes zoster virus (HZV)skin lesions, and also possibly inhibit both latent HSV infections and residual HZV infections.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active, latent or residual HSV or HZV infection

Exclusion Criteria:

* Unwilling or unable to provide Informed Consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HSV and HZV infected patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Expedited healing of active lesions | Within 1 day following therapy

SECONDARY OUTCOMES:
Recurrence of lesions and/or symptoms | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: W John Martin, MD, PhD, Principal Investigator — Institute of Progressive Medicine

REFERENCES:
- [Background] Martin WJ, Stoneburner J. Symptomatic relief of herpetic skin lesions utilizing an energy-based approach to healing. Exp Mol Pathol. 2005 Apr;78(2):131-4. doi: 10.1016/j.yexmp.2004.10.007. Epub 2005 Jan 5. PMID 15713438